CLINICAL TRIAL: NCT04816357
Title: Identification of Endometriosis and Migraine Criteria in Women With the Comorbidity of Both Conditions in Comparison With Women Who Only Suffer From Endometriosis - A Pilot Study
Status: Completed | Type: Observational
Sponsor: Zurich University of Applied Sciences (Other)
Responsible Party: Principal Investigator, Hanna Dietrich, Investigator, Zurich University of Applied Sciences
Other Study IDs: 2021-00285
Record Dates: First submitted 2021-03-22; First posted 2021-03-25 (Actual); Last update posted 2022-02-24 (Actual); Status verified 2022-02

CONDITIONS: Endometriosis; Migraine
MeSH Terms: conditions — Endometriosis; Migraine Disorders

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Endometriosis & Migraine: * Premenopausal women aged 18-55 years, at time of operation
  * Endometriosis confirmed with surgery and histologic staging (Report of the surgery available)
  * For the cases migraine needs to be confirmed during the interview according to the IHS criteria.
  Interventions: Other: Questionaire
- Endometriosis: * Premenopausal women aged 18-55 years, at time of operation
  * Endometriosis confirmed with surgery and histologic staging (Report of the surgery available)
  Interventions: Other: Questionaire

INTERVENTIONS:
Other: Questionaire — only questionaire

SUMMARY:
Patients with both, migraine and endometriosis, present the case-group, while women with endometriosis without migraine serve as controls. The primary endpoint is endometriosis stage confirmed by laparascopy compared to the control group. Further points to compare between groups are infertility, dysmenorrhea, dyschezia, dyspareunia, number of operations, family history with first-degree relatives, and age of first symptoms for both conditions and age at first operation.

Secondary endpoints to evaluate in percentages within the migraine group are migraine frequency, migraine aura/non-aura, age at migraine start, hormonal migraine, family history, treatment response, response to prophylactic agents, localization, types of aura and triggers. Other medical conditions and comorbidities like depression will be noted as well as response to Dienogest treatment.

In the questionnaire we will ask 62 Questions overall. The Questions for endometriosis are based on a questionnaire from the world endometriosis research foundation and to evaluate the severity of the migraine we will use the MIDAS (Migraine Disability Assessment) questionnaire (8).

ELIGIBILITY:
Inclusion Criteria:

* Premenopausal women aged 18-55 years, at time of operation
* Endometriosis confirmed with surgery and histologic staging (Report of the surgery available)
* For the cases migraine needs to be confirmed during the interview according to the IHS criteria.

Exclusion Criteria:

• Inability to perform the interview (insufficient knowledge of language, psychological disorder, dementia)

Ages: 18 Years to 99 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: From our database of operated endometriosis patients ranging from 2016-2020 100 women will be identified within the first phone call as cases with endometriosis and migraine and the threefold number (n=300) as control with endometriosis only.
Sampling Method: Probability Sample
Enrollment: 344 (Actual)
Dates: Start 2021-03-25 (Actual); Primary Completion 2021-11-04 (Actual); Study Completion 2021-11-04 (Actual)

PRIMARY OUTCOMES:
Endometriosis stage | 4 years
  endometriosis stage confirmed by laparascopy compared to the control group

SECONDARY OUTCOMES:
infertility, dysmenorrhea, dyschezia, dyspareunia, number of operations | 4 years
  s.o.
and age of first symptoms for both conditions and age at first operation | 4 years
  s.o.
family history with first-degree relatives, | 4 years
  s.o.
Secondary endpoints to evaluate in percentages within the migraine group are migraine frequency, migraine aura/non-aura, age at migraine start, hormonal migraine, family history, treatment response, | 4 years
  s.o.
response to prophylactic agents, localization, types of aura and triggers. Other medical conditions and comorbidities like depression will be noted | 4 years
  s.o.

CONTACTS AND LOCATIONS:
Locations (1):
- Universitätsspital Zürich, Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Dietrich H, Knobel C, Portmann L, Metzler J, Muendane A, Niggli A, Neumeier MS, Imesch P, Merki-Feld GS. Endometriosis features and dienogest tolerability in women with depression: a case-control study. Eur J Contracept Reprod Health Care. 2023 Jun;28(3):198-204. doi: 10.1080/13625187.2023.2199899. Epub 2023 May 3. PMID 37132337
- [Derived] Neumeier MS, Pohl H, Dietrich H, Knobel C, Portmann L, Metzler J, Imesch P, Merki-Feld GS. Endometriosis Features in Women With and Without Migraine. J Womens Health (Larchmt). 2023 May;32(5):598-607. doi: 10.1089/jwh.2022.0359. Epub 2023 Mar 10. PMID 36897310